CLINICAL TRIAL: NCT06738160
Title: The Efficacy and Safety of Narlumosbart in Combination With Stereotactic Body Radiation Therapy to Improve the Efficacy of First-line Chemotherapy Combined With Immunotherapy in Patients With Bone Metastases From Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-NSCLC-SBRT
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: NSCLC; Stereotactic Body Radiation Therapy (SBRT); Immunotherapy
MeSH Terms: interventions — Drug Therapy; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Narlumosbart (Experimental)
  Interventions: Drug: Narlumosbart

INTERVENTIONS:
Drug: Narlumosbart — Patients who have not received any systemic therapy will receive narlumosbart and bone target lesion SBRT in combination with first-line treatment immunotherapy and chemotherapy after screening eligible subjects. Narlumosbart, 120mg/time, subcutaneous injection, is administered every 4 weeks. For the treatment of SBRT for bone metastases, the dose of 24Gy/3F is used for spinal metastases, and 30Gy/5F or 35Gy/5F is used for non-spinal lesions. Chemotherapy combined with immune checkpoint inhibitor therapy was used in accordance with the guidelines. The primary endpoint is to assess the objective response rate of NSCLC patients with bone metastases from narlumosbart combined with SBRT and first-line chemotherapy and immunotherapy. The secondary endpoints include progression-free survival, overall survival and safety. Sample size calculation used the Simon Two-Stage method. 27 subjects will be enrolled in this project, considering the dropout rate of 10%.
  Other Names: chemotherapy; Stereotactic Body Radiation Therapy

SUMMARY:
Introduction: Immunotherapy in combination with chemotherapy have been recommended as the first-line treatment of driver-negative advanced non-small cell lung cancer (NSCLC), but the efficacy is worse in NSCLC patients with bone metastases due to the immunosuppressive microenvironment. Studies have shown that not only the nuclear factor kappa-B ligand (RANKL) inhibitors but also Stereotactic Body Radiation Therapy (SBRT) play a significant role in improving the tumor immune microenvironment. Therefore, narlumosbart，a monoclonal antibody (mAb) targeting RANKL，in combination with SBRT may have synergistic effects and improve efficacy of immunotherapy and chemotherapy in driver-negative advanced NSCLC patients with bone metastases.

Methods: This single-arm, single-center phase II clinical trial will enroll NSCLC patients with bone metastases who have not received any systemic therapy. Patients will receive narlumosbart and bone target lesion SBRT in combination with first-line treatment immunotherapy and chemotherapy after screening eligible subjects. Narlumosbart, 120mg/time, subcutaneous injection, is administered every 4 weeks. For the treatment of SBRT for bone metastases, the dose of 24Gy/3F is used for spinal metastases, and 30Gy/5F or 35Gy/5F is used for non-spinal lesions. Chemotherapy combined with immune checkpoint inhibitor therapy was used in accordance with the guidelines. The primary endpoint is to assess the objective response rate of NSCLC patients with bone metastases from narlumosbart combined with SBRT and first-line chemotherapy and immunotherapy. The secondary endpoints include progression-free survival, overall survival and safety. Sample size calculation used the Simon Two-Stage method. 9 patients will be enrolled in the first stage. If ≥ 2 patients achieve CR/PR, the second stage of enrollment will be performed. If only 2 patients < achieve CR/PR, the trial will be terminated. In the second phase, 15 patients will be enrolled. 27 subjects will be enrolled in this project, considering the dropout rate of 10%.

Wangjun Yan AND Zhengfei Zhu are the Co-Principal Investigators of this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to the implementation of any trial-related procedures;
* Age ≥ 18 years old and ≤ 80 years old;
* Histologically or cytologically confirmed stage IV NSCLC (International Association for the Study of Lung Cancer and American Joint Committee on Cancer Classification 9th Edition TNM Lung Cancer Staging);
* Histologically confirmed bone metastasis, which is assessed by the investigator to require local radiotherapy treatment;
* Patients who have not undergone systemic drug therapy for lung cancer (including chemotherapy, targeting, immunotherapy, etc.);
* Adenocarcinoma patients have been confirmed by tumour histology or cytology or haematology that the driver genes (EGFR, ALK, ROS-1) are all negative, and genetic testing is not required for squamous cell carcinoma patients;
* At least 1 evaluable lesion other than bone metastases (refer to RECIST1.1), and lymph nodes can be used as independent measurable lesions;
* Bone metastases other than the lesions to be radiotherapy do not require local treatment (surgery or radiotherapy) intervention after evaluation;
* ECOG score 0-1 points;
* Expected survival time > 3 months;
* Adequate organ function, subjects need to meet the following laboratory indicators: 1) In the absence of granulocyte colony-stimulating factor in the past 14 days, the absolute neutrophil value (ANC) ≥ 1.5x109/L; 2) In the case of no blood transfusion in the past 14 days, platelet ≥ 100×109/L; 3) In the absence of blood transfusion or erythropoietin in the past 14 days, haemoglobin > 9g/dL; 4) Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); 5) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) at 2.5 times ULN ≤ (subjects with liver metastases are allowed ALT or AST ≤5×ULN); 6) serum creatinine ≤ 1.5 times ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥ 60 ml/min; 7) good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; 8) Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within normal limits. If the baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled; 9) Cardiac enzyme spectrum within the normal range (if the investigator comprehensively judges that it is not clinically significant, simple laboratory abnormalities are also allowed to enroll); For female subjects of childbearing age, a urine or serum pregnancy test with a negative result should be received within 3 days prior to receiving the first dose of study drug (Cycle 1 Day 1). If the urine pregnancy test cannot be confirmed to be negative, a blood pregnancy test is required. Females of non-childbearing potential are defined as at least 1 year postmenopausal, or have undergone surgical sterilisation or hysterectomy; If there is a risk of conception, all participants, male or female, are required to use contraception with an annual failure rate of less than 1% throughout the treatment period until 120 days after the last dose of study drug (or 180 days after the last dose of study drug).

Exclusion Criteria:

* The pathology is small cell lung cancer (SCLC), including lung cancer mixed with SCLC and NSCLC;
* The lesion is an isolated lesion and can be treated radically;
* Patients who need surgical treatment after the evaluation of the study are not allowed to enroll;
* The radiotherapy lesion to be treated has been treated with radiotherapy or the lesion to be treated cannot be treated with radiotherapy after evaluation;
* Presence of active brain metastases;
* Diagnosis of other malignant diseases other than NSCLC within 5 years before the first dose (excluding radically cured basal cell carcinoma of the skin, squamous epithelial carcinoma of the skin, and/or carcinoma in situ after radical resection);
* Current participation in interventional clinical study treatment, or have received other investigational drugs or used investigational device treatment within 4 weeks prior to the first dose;
* Prior treatment with the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or targeting another stimulating or synergistic inhibition of T cell receptors (e.g., CTLA-4, OX-40, CD137) or targeting RANKL (denosumab, nalusolimab);
* Active autoimmune disease requiring systemic therapy (such as use of disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapies (e.g., thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
* Presence of clinically uncontrollable pleural effusion/ascites effusion (subjects who do not need to drain the effusion or stop draining for 3 days without significant increase in effusion can be enrolled);
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Presence of active bone metabolism disease (Paget bone disease, Cushing's syndrome, and hyperprolactinemia), rheumatoid arthritis, uncontrolled hyper/hypothyroidism, hyperparathyroidism/hypoparathyroidism;
* Those who are known to be allergic to the active ingredients or excipients such as sintilimab, pemetrexed, nalusopaimab, carboplatin, cisplatin, paclitaxel, etc., of the drug in this study;
* Have not recovered adequately from toxicity and/or complications induced by any of the interventions (i.e., ≤ grade 1 or to baseline, excluding fatigue or alopecia, prior to initiation of treatment);
* Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive);
* Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected at the same time greater than the upper limit of normal in the laboratory department of the research center);
* Hypocalcemia cannot be improved after treatment;
* Previous or current osteomyelitis or osteonecrosis of the jaw; Dental surgery or oral surgery that does not heal; Acute dental or jaw disease requiring oral surgery; Those who plan to undergo invasive dental surgery during the study;
* Use of any of the following anti-bone metabolizing agents within 6 months prior to enrollment: Parathyroid hormone (PTH) or derivatives; Calcitonin; Osteoprotein; Vaccination with a live vaccine within 30 days prior to the first dose (Cycle 1, Day 1);
* Pregnant or lactating women;
* Presence of any serious or uncontrollable systemic disease, such as:

  1. Resting ECG has major abnormalities in rhythm, conduction or morphology and severe symptoms that are difficult to control, such as complete left bundle branch block, heart block above degree II, ventricular arrhythmia or atrial fibrillation;
  2. unstable angina, congestive heart failure, New York Heart Association (NYHA) classification ≥ grade 2 chronic heart failure;
  3. myocardial infarction within 6 months prior to enrollment;
  4. unsatisfactory blood pressure control;
  5. History of non-infectious pneumonitis requiring glucocorticoid therapy within 1 year prior to the first dose, or current presence of clinically active interstitial lung disease;
  6. active tuberculosis;
  7. Presence of active or uncontrolled infection requiring systemic therapy;
  8. Presence of clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
  9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. poorly controlled diabetes mellitus (fasting blood glucose (FBG) >10mmol/L);
  11. Those whose urine routine showed a urine protein ≥++, and confirmed that the 24-hour urine protein was > 1.0 g;
  12. Subjects with mental disorders who are unable to cooperate with treatment; Medical history or evidence of disease, abnormal treatment or laboratory test values that may interfere with the results of the trial, prevent the subject from participating in the study throughout the study, or other conditions that are considered by the investigator to be unsuitable for enrollment in the opinion of the investigator are not suitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | 2 years

SECONDARY OUTCOMES:
Overall survival，OS | 2 years
  The time from enrollment to death from any cause. Patients who were still alive at the time of analysis will have the date of their last contact as the cutoff date.
Progression free survival, PFS | 2 years
  The time from enrollment to disease progression or death from any cause. Patients who were still alive at the time of analysis will have the date of their last contact as the cutoff date.
Adverse Events, AEs | 2 years
  AEs are crucial for assessing the safety profile of treatments in clinical trials and medical practice. The minimum Value is 0 ,indicating no occurrence of the adverse event. The maximum varies depending on the grading system used (e.g., Common Terminology Criteria for Adverse Events, CTCAE, which ranges from 1 to 5, with 5 indicating the most severe event, such as death.Higher scores indicate more severe adverse events. For example, in the CTCAE grading system: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death.
Brief Pain Inventory - Short Form, BPI-SF | 2 years
  Brief Pain Inventory - Short Form, BPI-SF is a widely used, self-administered questionnaire designed to assess the severity and impact of pain. The minimum value is 0 and the maximum value is 10. Higher scores indicate more severe pain or greater.Specifically, the BPI-SF includes assessments of pain intensity (e.g., worst pain, least pain, pain right now) and pain interference (e.g., interference with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life). Each item is rated on a scale from 0 (no pain or no interference) to 10 (worst possible pain or complete interference).
Skeletal-related event, SRE | 2 years
  Skeletal-related events (SREs) are complications that occur due to bone instability related to bone metastases or other bone-related diseases. The minimum value is 0, indicating no occurrence of skeletal-related events. The maximum value is not fixed, as the number and severity of SREs vary among individuals. A higher number and greater severity of SREs indicate more severe bone-related complications and worse clinical outcomes for the patient.
EORTC QLQ BM22 | 2 years
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Bone Metastases Module (EORTC QLQ-BM22) is a 22-item questionnaire specifically designed to assess the quality of life (QoL) in patients with bone metastases.Each item in the EORTC QLQ-BM22 is scored on a scale from 1 to 4, with the final scores being transformed into a standardized scale ranging from 0 to 100.For symptom scales, high score means worse outcomes. For function scales and psychosocial aspects, high score means better outcomes better functional ability and psychosocial well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China